CLINICAL TRIAL: NCT03474289
Title: A Phase 1 Study to Evaluate the Safety and Tolerability of SHR-1316 in Subjects With Advanced Tumors
Brief Title: Safety and Tolerability of SHR-1316 in Subjects With Advanced Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1316-I-101
Record Dates: First submitted 2018-03-11; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Escalation (Experimental): SHR-1316 administrated intravenously(IV) at protocol defined dose levels
  Interventions: Drug: SHR-1316
- Expansion (Experimental): SHR-1316 administrated IV in advanced solid tumors and selected tumor type
  Interventions: Drug: SHR-1316

INTERVENTIONS:
Drug: SHR-1316 — Monotherapy
  Other Names: HTI-1088

SUMMARY:
The purpose of this study is to access the safety and tolerability of the study drug known as SHR-1316 in metastatic/advanced malignancies

DETAILED DESCRIPTION:
This is an open-label, non-randomized, dose escalation/expansion phase I study, SHR-1316 is a humanized IgG4 monoclonal antibody that binds specifically to human PD-L1.The major aims of the study are to define the safety profile of this new drug, and to determine a recommended dose and schedule for potential additional trials.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age
2. Subjects with confirmed advanced malignancies (histologically or cytologically)
3. ECOG Performance status of 0 or 1
4. Adequate organ functions
5. Life expectancy ≥12 weeks;

Exclusion Criteria:

1. Subjects with active autoimmune disease.
2. Systemic cytotoxic chemotherapy, biological therapy, or major surgery within 4 weeks of the first dose of trial treatment
3. Previous received PD-1 or PD-L1 therapy
4. Known Active central nervous system (CNS) metastases
5. Known Clinically significant cardiovascular condition
6. Active infection or an unexplained fever >38.5°C
7. History of immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-01-30 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | at the end of cycle one(each cycle is 21 days)
  incidence and severity of treatment-related adverse events
Dose-limiting toxicities (DLTs) | at the end of cycle one(each cycle is 21 days)
  Number of participants with DLTs

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No